CLINICAL TRIAL: NCT01496716
Title: Obesity's Impact on the Clinical Efficacy and Quality of Life 1 Year After Primary Total Hip Arthroplasty
Brief Title: Obesity's Impact on the Effect of Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: THA-BMI
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Hip Osteoarthritis
Keywords: Osteoarthritis; obesity; quality of life
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Obesity | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip Osteoarthritis
  Interventions: Procedure: Hip arthroplasty

INTERVENTIONS:
Procedure: Hip arthroplasty — The purpose of hip arthroplasties is to reduce pain and increase mobility.

SUMMARY:
The purpose of this study is to investigate whether there is a correlation between hip arthroplasty patients' preoperative weight and the patients quality of life and the clinical effect one year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients recommended for primary total .

Exclusion Criteria:

* Rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hip total hip replacement patients operated on Hospital Southern Jutland, Denmark.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
SF-36 | Measured 1 week before surgery and 12 months postoperatively
  A patient reported outcome (PRO). The questionnaire is a tool for measuring health status. The form is used to measure the patient's view of his own health by scoring standardized responses to standardized questions. The schedule consists of 36 questions representing eight health concepts.

SECONDARY OUTCOMES:
HOOS | Measured 1 week before surgery and 12 months postoperatively
  Hip - specific patient-reported outcome that measures the patient's own assessment of hip problems and related problems. The schedule consists of 42 questions representing 5 strands.
Body composition | Measured 1 week before surgery and 12 months postoperatively
  Dual energy X-ray absorptiometry (DEXA) can measure total body bone mineral density and obtain accurate measurements of body tissue composition (muscle mass and fat mass). By measuring the body's muscle mass, fat mass and bone mineral density, one can estimate total body fat percentage.
Bone mineral density (BMD). | Measured 1 week before surgery and 12 months postoperatively
  Measured by DXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, professor, Principal Investigator — Department of Orthopedics Research Aarhus University Hospital
Locations (1):
- Department of Orthopedics Research Aarhus University Hospital, Aarhus C, Denmark